CLINICAL TRIAL: NCT06657209
Title: Normal-weight Diabetes: Adipocyte-directed Therapy with Pioglitazone or Tirzepatide
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tracey McLaughlin, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 77199
Record Dates: First submitted 2024-10-18; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test; Absorptiometry, Photon; Proton Magnetic Resonance Spectroscopy; Tirzepatide; Pioglitazone

STUDY DESIGN:
Intervention Model Description: Control group will undergo baseline testing to provide information about people without diabetes, but will not proceed with treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Normal weight controls (Other): Control
  Interventions: Procedure: Insulin resistance testing; Procedure: OGTT; Procedure: Fat biopsy; Radiation: DXA scan; Procedure: MRI; Procedure: 1H-MRS
- Normal weight with diabetes tirzepatide first pioglitazone second (Experimental): Baseline testing Intervention with tirzepatide for 16 weeks Retesting Washout for 5 weeks Intervention with pioglitazone for 16 weeks Retesting
  Interventions: Procedure: Insulin resistance testing; Procedure: OGTT; Procedure: Fat biopsy; Radiation: DXA scan; Procedure: MRI; Procedure: 1H-MRS; Drug: Tirzepatide; Drug: Pioglitazone
- Normal weight with diabetes pioglitazone first, tirzepatide second (Experimental): Baseline testing Intervention with pioglitazone for 16 weeks Retesting Washout for 5 weeks Intervention with tirzepatide for 16 weeks Retesting
  Interventions: Procedure: Insulin resistance testing; Procedure: OGTT; Procedure: Fat biopsy; Radiation: DXA scan; Procedure: MRI; Procedure: 1H-MRS; Drug: Tirzepatide; Drug: Pioglitazone

INTERVENTIONS:
Procedure: Insulin resistance testing — Steady state Plasma Glucose test
  Other Names: SSPG
Procedure: OGTT — Will collect 5 blood draws during the test to measure insulin secretion
  Other Names: Oral glucose tolerance test
Procedure: Fat biopsy — Needle biopsy to gather a sample of abdominal subcutaneous fat
Radiation: DXA scan — Whole body DXA scan
Procedure: MRI — Abdominal MRI
Procedure: 1H-MRS — Spectroscopy of the abdominal region
  Other Names: proton magnetic resonance spectroscopy
Drug: Tirzepatide — 16 weeks started at 2.5mg/week and increased to 5mg/week dose
  Other Names: Mounjaro
  Arms: Normal weight with diabetes pioglitazone first, tirzepatide second; Normal weight with diabetes tirzepatide first pioglitazone second
Drug: Pioglitazone — 16 weeks at a 45mg/day dose
  Other Names: Actos
  Arms: Normal weight with diabetes pioglitazone first, tirzepatide second; Normal weight with diabetes tirzepatide first pioglitazone second

SUMMARY:
This study is to investigate how adipocyte (fat cell) function and fat distribution differ between individuals with normal-weight type 2 diabetes (NWD) and normal-weight controls without diabetes (NWC). The study will assess whether adipocyte-directed therapies, specifically pioglitazone and tirzepatide, can improve insulin resistance, adipocyte function, and fat distribution in individuals with NWD. By analyzing the biological mechanisms underlying adipocyte dysfunction, the study aims to provide insights into novel treatment strategies for improving metabolic health in normal-weight individuals with type 2 diabetes.

DETAILED DESCRIPTION:
The investigators aim to learn how adipocyte dysfunction and disordered fat distribution contribute to the development of type 2 diabetes in normal-weight individuals. The investigators hope to determine whether adipocyte-directed therapies, such as pioglitazone and tirzepatide, can improve insulin sensitivity, fat distribution, and metabolic health in this population. This study is important because most diabetes research focuses on overweight or obese individuals, and very little is known about how diabetes affects those with normal body weight. Understanding the unique biology of normal-weight diabetes could lead to more personalized and effective treatment strategies, filling a gap in diabetes care for a group that can be overlooked in clinical research.

ELIGIBILITY:
Inclusion Criteria:

Normal-Weight Diabetes (NWD) Group:

1. Age: 30 to 70 years old.
2. Diagnosis of Type 2 Diabetes (T2D): Based on a previous diagnosis or confirmed by laboratory testing at screening (A1c > 5.7% or fasting glucose > 100 mg/dL).
3. HbA1c Range: Between 5.7% and 8%, with a stable medication or lifestyle regimen for at least 3 months.
4. BMI: Between 19 and 24.9 kg/m².
5. Diabetes Medications: All diabetes medications are allowed, except insulin and pioglitazone. GLP-1 receptor agonists are permitted if the dose has been stable for 3 months.
6. Stable Body Weight: Body weight must have been stable (no more than 2 kg change) over the last 3 months.

Normal-Weight Control (NWC) Group:

1. Age: 30 to 70 years old.
2. No Diagnosis of Diabetes: Fasting plasma glucose < 100 mg/dL and A1c < 5.7%, with no history of glucose-lowering medications.
3. BMI: Between 19 and 24.9 kg/m².
4. Stable Body Weight: No more than 2 kg change over the past 3 months. -

Exclusion Criteria:

1. Pregnancy or Lactation: Women who are pregnant, planning to become pregnant, or breastfeeding are excluded due to potential risks to the fetus or infant.
2. Prior Use of Pioglitazone: Participants who have previously used pioglitazone are excluded to avoid confounding effects of prior drug exposure.
3. Unstable Body Weight: Individuals with a body weight change of more than 2 kg in the last 3 months are excluded to ensure stable metabolic conditions.
4. Liver or Kidney Disease: Participants with significant liver disease (ALT > 3x upper limit of normal) or renal disease (creatinine > 1.5 mg/dL) are excluded due to potential safety risks.
5. Congestive Heart Failure or Fluid Overload History: These conditions are exclusionary due to the risk of fluid retention with pioglitazone.
6. Uncontrolled Hypertension: Blood pressure > 160/90 mmHg excludes participants due to increased cardiovascular risk.
7. Active Cancer: Individuals with a diagnosis of cancer in the past 3 years (except for skin cancer) are excluded.
8. Chronic Inflammatory Diseases: Excluded due to potential effects on metabolic measurements.
9. Use of Weight Loss Medications: Those currently taking weight loss medications are excluded to prevent confounding effects on body weight and metabolic function.
10. Bariatric Surgery or Liposuction History: Participants who have had weight-loss surgeries or liposuction are excluded due to alterations in fat tissue and metabolic profiles.
11. Insulin Use: Participants using insulin are excluded to focus on non-insulin-dependent diabetes.
12. Active Psychiatric Disease or Eating Disorders: Individuals with these conditions are excluded due to potential impacts on study compliance and data integrity.
13. Substance Abuse: Participants with a history of substance abuse are excluded for similar reasons.

    -

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance in normal weight women with diabetes compared to those with no diabetes | Baseline measures comparison between the groups
  Insulin resistance will be measured by a Steady State Plasma Glucose test (SSPG). Results will be measured by glucose levels at steady state in mg/dL.
Adipocyte function in women with normal weight diabetes as compared with those without diabetes | Baseline comparisons
  Adipocyte function will be measured as percent small adipocytes and peak diameter adipocytes from the fat biopsies.
Fat storage in women with normal weight diabetes compared to those without diabetes | Baseline comparisons between the groups
  Fat storage will be measured by MRI. Quantification of subcutaneous and visceral abdominal fat will be obtained by MRI using a fat-water imaging sequence (parameters: IDEAL-IQ: 3D GRE, 160x160 matrix, 6 echoes, 4 degree flip angle, minimum TR = 7.3 ms, 28 slices, 10 mm slice thickness.

SECONDARY OUTCOMES:
Effect of adipose-directed therapy pioglitazone on HbA1c in both men and women with normal weight diabetes | 16 weeks
  Hemoglobin A1C measures will be compared baseline to end of 16 weeks of intervention with pioglitazone.
Effect of pioglitazone in insulin resistance in both men and women. | 16 weeks
  SSPG test results will be compared from baseline to end of pioglitazone intervention.
  Results will be measured by glucose levels at steady state in mg/dL.
Fat storage in men with normal weight diabetes (NWD) compared to those without diabetes (NWC). | Baseline comparisons between the groups
  Fat storage will be measured by MRI. Quantification of subcutaneous and visceral abdominal fat will be obtained by MRI using a fat-water imaging sequence (parameters: IDEAL-IQ: 3D GRE, 160x160 matrix, 6 echoes, 4 degree flip angle, minimum TR = 7.3 ms, 28 slices, 10 mm slice thickness.
Adipocyte function in men with normal weight diabetes as compared with those without diabetes | Baseline comparisons
  Adipocyte function as measured by percent small adipocytes and peak diameter adipocytes from the fat biopsies.
Insulin resistance in normal weight men with diabetes compared to those with no diabetes | Baseline measures comparison between the groups
  Insulin resistance will be measured by a Steady State Plasma Glucose test (SSPG). Results will be measured by glucose levels at steady state in mg/dL.
Insulin secretion in men and women with normal weight diabetes compared to those without diabetes | Baseline measured compared between the groups
  A five-point, three-hour OGTT will be done after overnight fast for calculation of insulin secretion using c-peptide deconvolution, and disposition index calculated by dividing this value by SSPG.

OTHER OUTCOMES:
Effect of adipose-directed therapy with tirzepatide on insulin resistance in men and women with normal weight diabetes (NWD). | 16 weeks
  SSPG test results will be compared from baseline to end of tirzepatide intervention. Results will be measured by glucose levels at steady state in mg/dL.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Clinical and Translational Research Unit (CTRU), Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No